CLINICAL TRIAL: NCT00703976
Title: Phase II Randomized Trial of Radiation, Cetuximab and Pemetrexed With or Without Bevacizumab in Locally Advanced Head and Neck Cancer
Brief Title: Radiation, Cetuximab and Pemetrexed With or Without Bevacizumab in Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eli Lilly and Company (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-021
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Cancer
Keywords: head and neck cancers
MeSH Terms: conditions — Neoplasms; Head and Neck Neoplasms | interventions — Bevacizumab; Cetuximab; Pemetrexed; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab, Pemetrexed and Radiation therapy (Active Comparator): Cetuximab, Pemetrexed and Radiation therapy Cetuximab: Cetuximab is approved by the FDA for head and neck cancers in patients who have failed other chemotherapy treatments.
  Pemetrexed: Pemetrexed is approved by the Food and Drug Administration (FDA) for head and neck cancer when used in combination with radiation therapy.
  Radiation therapy: Radiation therapy standard fractionation 2 Gy/day without planned interruptions beginning on day 1 (Monday or Tuesday preferred). Radiation will be given 5 days/week, Monday through Friday, for 7 consecutive weeks
  Interventions: Drug: Cetuximab; Drug: Pemetrexed; Radiation: Radiation therapy
- Cetuximab, Pemetrexed, Radiation Therapy plus Bevacizumab (Experimental): Cetuximab, Pemetrexed, Radiation Therapy plus Bevacizumab Cetuximab: Cetuximab is approved by the FDA for head and neck cancers in patients who have failed other chemotherapy treatments.
  Pemetrexed: Pemetrexed is approved by the Food and Drug Administration (FDA) for head and neck cancer when used in combination with radiation therapy.
  Radiation therapy: Radiation therapy standard fractionation 2 Gy/day without planned interruptions beginning on day 1 (Monday or Tuesday preferred). Radiation will be given 5 days/week, Monday through Friday, for 7 consecutive weeks Bevacizumab: Bevacizumab is approved by the Food and Drug Administration (FDA) for colorectal cancer and non-small cell lung cancer in combination of chemotherapy.
  Interventions: Drug: Bevacizumab; Drug: Cetuximab; Drug: Pemetrexed; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab is approved by the Food and Drug Administration (FDA) for colorectal cancer and non-small cell lung cancer in combination of chemotherapy.
  Other Names: Avastin
  Arms: Cetuximab, Pemetrexed, Radiation Therapy plus Bevacizumab
Drug: Cetuximab — Cetuximab is approved by the FDA for head and neck cancers in patients who have failed other chemotherapy treatments.
  Other Names: Erbitux
Drug: Pemetrexed — Pemetrexed is approved by the Food and Drug Administration (FDA) for head and neck cancer when used in combination with radiation therapy.
  Other Names: Alimta
Radiation: Radiation therapy — Radiation therapy standard fractionation 2 Gy/day without planned interruptions beginning on day 1 (Monday or Tuesday preferred). Radiation will be given 5 days/week, Monday through Friday, for 7 consecutive weeks

SUMMARY:
The purpose of this study is to compare the effects (good and bad) of chemoradiotherapy with or without Bevacizumab (Avastin). Chemoradiotherapy is the combination of chemotherapy (the drugs pemetrexed and cetuximab) and radiation. Pemetrexed is not approved by the Food and Drug Administration (FDA) for head and neck cancer when used in combination with radiation therapy. Cetuximab is also approved by the FDA for head and neck cancers in patients who have failed other chemotherapy treatments. Bevacizumab is approved by the Food and Drug Administration (FDA) for colorectal cancer and non-small cell lung cancer in combination of chemotherapy. In this study, the use of bevacizumab is investigational.

DETAILED DESCRIPTION:
Background

Patients with squamous cell carcinoma of the head and neck (HNSCC) are increasingly treated with primary chemoradiotherapy. The incorporation of novel targeted therapies to chemoradiotherapy is of major interest since it may potentially improve efficacy without significantly increasing toxicity. Radiation and cetuximab, a chimeric anti-epidermal growth factor receptor monoclonal antibody, has emerged as a standard non-surgical therapy for stage III/IV HNSCC. Bevacizumab, an anti-vascular endothelial growth factor antibody is currently being investigated in HNSCC with promising results. A phase II study investigating the combination of pemetrexed and bevacizumab in recurrent or metastatic HNSCC is currently ongoing at our institution with encouraging results (UPCI# 05-002). In addition, we are completing a phase I trial of radiation, cetuximab plus pemetrexed (UPCI #05-005). Pemetrexed was dose escalated in successive cohorts of patients on 3 dose levels: starting dose level (0) 350 mg/m2, dose level (-1) 200 mg/m2, dose level (+1) 500 mg/m2. Currently three patients have been treated at dose level +1 (pemetrexed 500 mg/m2) which will be the pemetrexed dose in this study. No dose limiting toxicities (DLTs) have been observed at this dose level, which was the maximum tolerated dose (MTD) for the combination regimen in previously non-irradiated patients.

Specific aims

To evaluate the progression-free survival at 2 years (primary endpoint), locoregional and distant disease-free survival, overall survival, toxicities and quality of life with the combination of radiation, cetuximab and pemetrexed with or without bevacizumab in patients with locally advanced HNSCC. Also, we plan to collect tumor tissue from previous diagnostic procedures and baseline blood specimens for future correlative studies.

Subject population

We will enroll patients with previously untreated stage III/IV squamous cell carcinoma or undifferentiated carcinoma of the head and neck (except nasopharynx and unknown primary). Patients should not have active bleeding due to HNSCC or history of persistent bleeding due to HNSCC that required major intervention (surgery or embolization) to be controlled. Please see section 3 for detailed eligibility criteria.

Treatment plan

Patients will be randomized in two arms. In arm A, patients will be treated with radiation 2Gy/day for 7 weeks to a total of 70 Gy, cetuximab 250mg/m2 weekly during radiation, after a loading dose of 400mg/m2 one week prior starting radiation, and pemetrexed 500mg/m2 every 21 days for 3 cycles. In arm B, patients will be treated with the same regimen with the addition of bevacizumab 15mg/kg every 21 days for 3 cycles (see section 5 for detailed treatment plan and dose modifications).

Statistical design and sample size

Phase II, randomized, multi-center study with progression-free survival at 2 years as the primary endpoint. The historical control is a 2-year progression-free survival of 46% with radiation plus cetuximab alone. We assume a 2 year progression free survival of 64% (40% relative improvement in progression-free survival over historical control) as worthy of further testing. We will require 40 evaluable patients per arm for a total of 80 patients. Alpha = 0.1, beta = 0.1; all tests one-tailed.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have pathologically confirmed AJCC 6th edition (see Appendix) stage III or IV (M0) squamous cell carcinoma or undifferentiated or poorly differentiated carcinoma of the oropharynx, larynx, or hypopharynx with no evidence of distant metastasis. Biopsy sampling of primary tumor with pathology report documentation of confirmed diagnostic tissue type is required. Patients should be evaluated by a Radiation Oncologist, Medical Oncologist and Otolaryngologist prior to enrolling on study.
* No prior treatment for head and neck cancer. Limited, organ-preserving surgery is allowed
* ECOG performance status 0-1
* Unidimensionally measurable disease is not required. However, patients should require treatment with full dose radiotherapy (not postoperative)
* Age greater or equal to 18 years
* Absolute neutrophil count greater or equal to 1500/µl, Platelet count greater or equal to 100,000/µl
* Creatinine clearance 45 ml/min or higher calculated using the Cockcroft-Gault formula
* Total bilirubin within normal limits and AST/ALT less than 3 times the upper limit of normal
* Urine protein should be screened by urine analysis for Urine Protein Creatinine (UPC) ratio. For UPC ratio >0.5, 24-hour urine protein should be obtained and the level must be <1000mg for patients to be eligible
* Informed consent must be obtained from all patients prior to beginning therapy. Patients should have the ability to understand and the willingness to sign a written informed consent document
* Patients should be willing and able to take folic acid and vitamin B12 supplementation and should interrupt aspirin or other non-steroidal anti-inflammatory agents for a 5-day period
* The use of anti-platelet agents(e.g. dipyridamole (Persatine), ticlopidine (Ticlid), clopidogrel (Plavix)) is allowed only if patient is not receiving aspirin or NSAID's known to inhibit platelet function.
* Patients who meet the following criteria will be excluded due to the possibility of increased risk for tumor bleeding with bevacizumab therapy:

  * active bleeding due to head and neck cancer of more than ½ teaspoon of bright red blood per episode or history of persistent bleeding due to SCCHN that required major intervention (surgery or embolization) to be controlled.
  * history of gross hemoptysis (bright red blood of .05 teaspoon or more per episode of coughing) less than or equal to 3 months prior to enrollment
  * history of coagulopathy or hemorrhagic disorders
* Patients should not be on therapeutic anticoagulation (prophylactic use of warfarin 1 mg per day is allowed) and INR should be < 1.5 at registration.
* Patients with a prior history of squamous cell or basal carcinoma of the skin or in situ cervical cancer must have been curatively treated. Patients with a history of other prior malignancy must have been treated with curative intent and must have remained disease-free for 5 years post diagnosis
* Patients with history of hypertension must be well-controlled upon study entry (≤150/90) on a stable regimen of anti-hypertensive therapy. Patients should not have any prior history of hypertensive crisis or hypertensive encephalopathy.
* No major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment, or anticipation of need for major surgical procedure during the course of the study. Prior surgical therapy will consist only of incisional or excisional biopsy and organ sparing procedures such as debulking of airway compromising tumors or neck dissection in a patient with an existing primary tumor. Any non-biopsy procedure must have taken place >4 weeks but <3 months of initiating protocol treatment. No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to registration. No serious non-healing wound, ulcer, or bone fracture.
* No unstable angina or myocardial infarction within the previous 6 months; no symptomatic congestive heart failure; no serious cardiac arrhythmia requiring medication; no clinically significant peripheral vascular disease; no history of aortic dissection; no history of any CNS cerebrovascular ischemia or stroke within the last 6 months; no active serious infection. All patients will have a baseline EKG. If abnormalities consistent with active coronary artery disease are detected, the patient will be referred to a cardiologist for appropriate evaluation and management prior to treatment on study
* For patients who have baseline clinically significant pleural or peritoneal effusions (on the basis of symptoms or clinical examination) before initiation of protocol therapy, consideration should be given to draining the effusion prior to starting therapy due the potential of increased toxicity with pemetrexed in that setting
* Submission of archival tumor samples, unstained slides or blocks, for correlative studies is strongly encouraged, but not required for subject participation if tissue is not readily available or quantity is not sufficient for release per submitting pathologist.

Exclusion Criteria:

* Patients who are receiving any other investigational agents.
* Ineligible will be patients with uncontrolled intercurrent illness including, but not limited to,ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients should not have prior history of a serious reaction to a monoclonal antibody. Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies are not eligible.
* Women must not be pregnant or breast feeding because chemotherapy may be harmful to the fetus or the nursing infant. Pregnant women are excluded from this study because chemotherapy and/or bevacizumab have the potential for teratogenic or abortifacient effects.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible drug interactions with study drugs. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Bauman, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 80 patients were enrolled, only 78 began the study because 2 were found to be ineligible prior to treatment.
Period: Overall Study
Arm/Group | Cetuximab, Pemetrexed and Radiation Therapy | Cetuximab, Pemetrexed, Radiation Therapy Plus Bevacizumab
Started | 37 | 41
Completed | 37 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab, Pemetrexed and Radiation Therapy | Cetuximab, Pemetrexed, Radiation Therapy Plus Bevacizumab | Total
Number analyzed (Participants) | 37 | 41 | 78
Age, Continuous [Median (Full Range); unit: years] | 57 [39 to 69] | 56 [35 to 76] | 56 [35 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 32 | 31 | 63

OUTCOME MEASURES:

1. Primary Outcome: 2-year Progression-free Survival (PFS)
Description: Two-year PFS is an estimated percentage of participants without disease progression (locoregional or distant) at two years after the start of study treatment. Progression was defined using Response Evaluation Criteria In Solid Tumors (RECIST v1.0), as: at least a 20% (and at least 5 millimeters) increase in the sum of the diameters of target lesions, or the appearance of one or more new lesions.
Time Frame: 18 months to patient accrual and 2 years of follow-up after closing accrual.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab, Pemetrexed and Radiation Therapy | Cetuximab, Pemetrexed, Radiation Therapy Plus Bevacizumab
Number analyzed (Participants) | 37 | 41
percentage of participants | 79 [69 to 92] | 75 [64 to 88]

2. Secondary Outcome: 2-year Overall Survival (OS)
Description: Two-year OS is an estimated percentage of participants still living at two years after the start of study treatment.
Time Frame: 2 years of follow-up after closing accrual
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants (Overall Study) | Cetuximab, Pemetrexed and Radiation Therapy | Cetuximab, Pemetrexed, Radiation Therapy Plus Bevacizumab
Number analyzed (Participants) | 78 | 37 | 41
percentage of participants | 88 [81 to 96] | 91 [82 to 100] | 87 [77 to 98]

ADVERSE EVENTS:
Description: Adverse events were not collected/monitored "per Arm/Group"
Arm/Group | All Participants (Overall Study)
Serious Adverse Events (participants affected / at risk) | 31/78
Other Adverse Events (participants affected / at risk) | 78/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (Overall Study) (N=78)
Hemoglobin (Blood and lymphatic system disorders) | 1
Leukocytes (total WBC) (Investigations) | 1
Lymphopenia (Investigations) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2
Hypotension (Vascular disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2
Weight loss (Investigations) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Rash: dermatitis associated with radiation, Chemoradiation (Skin and subcutaneous tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 4
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2
Gastrointestinal - Other (Gastrointestinal disorders) | 2
Leak (including anastomotic), GI, Leak NOS (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 6
Mucositis/stomatitis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1
Ulcer, GI, Stomach (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Hemorrhage, GI, Oral cavity (Gastrointestinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory, Pharynx (Respiratory, thoracic and mediastinal disorders) | 1
Febrile neutropenia (fever of unknown origin without documented infection) (Blood and lymphatic system disorders) | 2
Infection - Other (Infections and infestations) | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L), Skin (cellulitis) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Lung (pneumonia) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Meninges (meningitis) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Skin (cellulitis) (Infections and infestations) | 1
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1
Confusion (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 2
Syncope (fainting) (Nervous system disorders) | 1
Pain, Abdomen NOS (Gastrointestinal disorders) | 2
Pain, Head/headache (Nervous system disorders) | 1
Pain, Oral cavity (Gastrointestinal disorders) | 6
Pain, Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (Overall Study) (N=78)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Auditory/Ear - Other (Ear and labyrinth disorders) | 3
Otitis, external ear (non-infectious) (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 4
Haptoglobin (Investigations) | 1
Hemoglobin (Blood and lymphatic system disorders) | 55
Leukocytes (total WBC) (Investigations) | 59
Lymphopenia (Investigations) | 61
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 50
Platelets (Investigations) | 25
Supraventricular and nodal arrhythmia, Sinus bradycardia (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia, Sinus tachycardia (Cardiac disorders) | 2
Cardiac General - Other (Cardiac disorders) | 4
Hypertension (Vascular disorders) | 12
Hypotension (Vascular disorders) | 7
Coagulation - Other (Blood and lymphatic system disorders) | 1
INR (International Normalized Ratio of prothrombin time) (Vascular disorders) | 6
PTT (Partial Thromboplastin Time) (Vascular disorders) | 3
Constitutional Symptoms - Other (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 57
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 20
Insomnia (Psychiatric disorders) | 19
Rigors/chills (General disorders) | 13
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1
Weight loss (Investigations) | 50
Burn (Injury, poisoning and procedural complications) | 3
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 21
Dry skin (Skin and subcutaneous tissue disorders) | 44
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 6
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Injection site reaction/extravasation changes (General disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 13
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 55
Rash: dermatitis associated with radiation, Chemoradiation (Skin and subcutaneous tissue disorders) | 33
Rash: dermatitis associated with radiation, Radiation (Skin and subcutaneous tissue disorders) | 52
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 4
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Ulceration (General disorders) | 11
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1
Endocrine - Other (Endocrine disorders) | 1
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 3
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 16
Constipation (Gastrointestinal disorders) | 36
Dehydration (Metabolism and nutrition disorders) | 21
Dental: dentures or prosthesis (Gastrointestinal disorders) | 2
Dental: teeth (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 16
Distension/bloating, abdominal (Gastrointestinal disorders) | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 52
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 56
Esophagitis (Gastrointestinal disorders) | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 16
Heartburn/dyspepsia (Gastrointestinal disorders) | 17
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam), Larynx (Respiratory, thoracic and mediastinal disorders) | 1
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 36
Mucositis/stomatitis (clinical exam), Pharynx (Respiratory, thoracic and mediastinal disorders) | 1
Mucositis/stomatitis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 48
Mucositis/stomatitis (functional/symptomatic), Pharynx (Respiratory, thoracic and mediastinal disorders) | 2
Nausea (Gastrointestinal disorders) | 45
Perforation, GI, Colon (Gastrointestinal disorders) | 1
Salivary gland changes/saliva (Gastrointestinal disorders) | 25
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 36
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 1
Ulcer, GI, Duodenum (Gastrointestinal disorders) | 1
Ulcer, GI, Stomach (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 26
Hemorrhage, GI, Anus (Gastrointestinal disorders) | 1
Hemorrhage, GI, Oral cavity (Gastrointestinal disorders) | 1
Hemorrhage, GU, Urinary NOS (Renal and urinary disorders) | 3
Hemorrhage, pulmonary/upper respiratory, Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory, Nose (Respiratory, thoracic and mediastinal disorders) | 11
Hemorrhage, pulmonary/upper respiratory, Pharynx (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory, Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage/Bleeding - Other (Blood and lymphatic system disorders) | 8
Febrile neutropenia (fever of unknown origin without documented infection) (Blood and lymphatic system disorders) | 2
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L), Neck NOS (Infections and infestations) | 1
Infection - Other (Infections and infestations) | 35
Infection with normal ANC or Grade 1 or 2 neutrophils, Abdomen NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Foreign body (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils, Lung (pneumonia) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Neck NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Oral cavity-gums (gingivitis) (Infections and infestations) | 3
Infection with normal ANC or Grade 1 or 2 neutrophils, Upper aerodigestive NOS (Infections and infestations) | 1
Infection with unknown ANC, Dental-tooth (Infections and infestations) | 1
Infection with unknown ANC, Foreign body (e.g., graft, implant, prosthesis, stent) (Infections and infestations) | 1
Infection with unknown ANC, Neck NOS (Infections and infestations) | 1
Infection with unknown ANC, Skin (cellulitis) (Infections and infestations) | 2
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 1
Edema: head and neck (General disorders) | 10
Edema: limb (General disorders) | 3
Lymphatics - Other (Blood and lymphatic system disorders) | 4
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 37
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 35
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 55
Alkaline phosphatase (Investigations) | 13
Bicarbonate, serum-low (Investigations) | 3
Bilirubin (hyperbilirubinemia) (Investigations) | 6
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 8
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 35
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 3
Creatinine (Investigations) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 60
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 5
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 18
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 17
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 23
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 16
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 16
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 19
Proteinuria (Renal and urinary disorders) | 5
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 3
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 50
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1
Cervical spine-range of motion (Musculoskeletal and connective tissue disorders) | 1
Fibrosis-deep connective tissue (Musculoskeletal and connective tissue disorders) | 6
Fracture (Injury, poisoning and procedural complications) | 1
Joint-function (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness, generalized or specific area (not due to neuropathy), Extremity-upper (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy), Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 16
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Soft tissue necrosis, Neck (Musculoskeletal and connective tissue disorders) | 1
Trismus (difficulty, restriction or pain when opening mouth) (Musculoskeletal and connective tissue disorders) | 12
Cognitive disturbance (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 3
Dizziness (Nervous system disorders) | 9
Memory impairment (Nervous system disorders) | 3
Mental status (Psychiatric disorders) | 2
Mood alteration, Agitation (Psychiatric disorders) | 1
Mood alteration, Anxiety (Psychiatric disorders) | 11
Mood alteration, Depression (Psychiatric disorders) | 8
Neurology - Other (Nervous system disorders) | 2
Neuropathy: sensory (Nervous system disorders) | 3
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1
Seizure (Nervous system disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 3
Dry eye syndrome (Eye disorders) | 1
Vision-blurred vision (Eye disorders) | 2
Vision-flashing lights/floaters (Eye disorders) | 1
Vision-photophobia (Eye disorders) | 2
Watery eye (epiphora, tearing) (Eye disorders) | 1
Pain - Other (General disorders) | 44
Pain, Abdomen NOS (Gastrointestinal disorders) | 2
Pain, Back (Musculoskeletal and connective tissue disorders) | 2
Pain, Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 2
Pain, Dental/teeth/peridontal (Gastrointestinal disorders) | 1
Pain, Esophagus (Gastrointestinal disorders) | 3
Pain, External ear (Ear and labyrinth disorders) | 2
Pain, Extremity-limb (Musculoskeletal and connective tissue disorders) | 3
Pain, Face (General disorders) | 3
Pain, Head/headache (Nervous system disorders) | 28
Pain, Joint (Musculoskeletal and connective tissue disorders) | 1
Pain, Larynx (Respiratory, thoracic and mediastinal disorders) | 2
Pain, Muscle (Musculoskeletal and connective tissue disorders) | 1
Pain, Neck (Musculoskeletal and connective tissue disorders) | 14
Pain, Oral cavity (Gastrointestinal disorders) | 20
Pain, Pain NOS (General disorders) | 16
Pain, Skin (Skin and subcutaneous tissue disorders) | 1
Pain, Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 35
Pain, Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 7
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 30
Renal/Genitourinary - Other (Renal and urinary disorders) | 3
Erectile dysfunction (Reproductive system and breast disorders) | 1
Libido (Reproductive system and breast disorders) | 1
Sexual/Reproductive Function - Other (Reproductive system and breast disorders) | 1
Flu-like syndrome (General disorders) | 1
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
Vascular - Other (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes